CLINICAL TRIAL: NCT04087356
Title: Age-related Macular Degeneration (AMD) and Cardiovascular Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The New York Eye & Ear Infirmary (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-19-01872
Record Dates: First submitted 2019-07-09; First posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Age-related Macular Degeneration; Coronary Artery Disease; Cardiovascular Diseases
MeSH Terms: conditions — Macular Degeneration; Coronary Artery Disease; Cardiovascular Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood draw for serum markers and genetics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RMD+ Patients: Age-related macular degeneration patients with reticular macular disease
  Interventions: Genetic: Blood draw
- RMD- Patients: Age-related macular degeneration patients without reticular macular disease
  Interventions: Genetic: Blood draw

INTERVENTIONS:
Genetic: Blood draw — Blood samples are collected for genetic analysis, looking specifically at serum lipids and the inflammatory biomarker hs-CRP.

SUMMARY:
The purpose of this research study is to investigate the link between age-related macular degeneration (AMD or ARMD) and coronary artery disease (CAD). Age-related macular degeneration is a medical condition which may result in blurred or no vision in the center of vision. Coronary artery disease is a blockage of one or more arteries that supply blood to the heart. The study will specifically look at the macular changes that occur in the retina, which is the sensory membrane that lines the inner surface at the back of the eyeball, and the relationship between coronary heart disease and the risk factors.

DETAILED DESCRIPTION:
The treatment of age-related macular degeneration (AMD), the leading cause of blindness in the developed world, is undergoing a revolution. Intraocular injections of medications that can shut down the rapidly destructive "wet" form of the disease have changed this form to a chronic illness. However, vision is still lost. For the early forms of AMD, progression to the advanced "wet" and "dry" forms and severe vision loss is impeded but not stopped by current therapies of oral antioxidants. Thus, a better understanding of early AMD is needed to discover its root causes and provide treatment before irreparable damage is done.

The most important, highest-risk, and least understood form of early AMD is "reticular macular disease" (RMD). RMD is associated with significant progression to advanced AMD, both wet and dry. The lesions of RMD are well seen on the advanced retinal imaging techniques of spectral domain optical coherence tomography (SD-OCT) and scanning laser ophthalmoscopy (SLO). On SLO, RMD presents a pox-like pattern of dark defects SD-OCT provides high-resolution cross-sectional images of the retina, where RMD is seen as a collection of cholesterol-containing deposits, and the choroid, an essential blood supply of the retina, which is thinned and may be damaged in RMD. A unified explanation of these facets of RMD is lacking.

Regarding AMD and systemic diseases, the association between stroke, heart attack and AMD has been studied, but with some conflicting findings. For example, a relationship with heart attack has been established in patients less than age 75, but not in older patients. Where does RMD fit in? At present, no one knows. However, the known facts are these: RMD is associated with decreased longevity, which is not the case with other early forms of AMD. This could happen if RMD and systemic vascular disease co-exist. Finally, there is the very high proportion of women relative to men among older patients with RMD, about 85%. Women develop heart disease later than men and survive heart disease a decade longer on average. It is possible that these diseases both begin earlier in life, with more men dying before reaching older ages and demonstrating RMD. The research team submitting this proposal has preliminary data suggesting that this is in fact the case.

In a small group of subjects 50-75 years old, RMD was detected in a significant proportion of those with CAD compared to those without. Furthermore, in this younger group, the ratio of men to women in the RMD group was equal. The team proposes a large-scale initiative to provide definitive answers to these questions, in collaboration with expert cardiologists and neurologists to document vascular status unequivocally, and utilizing the most advanced retinal imaging available for the detection of RMD. This could lead to greater understanding of all three, stroke, heart attack and AMD, and ultimately better treatment, providing much needed relief to suffering patients and relief to the healthcare burden of an aging population.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of age-related macular degeneration in at least one eye.
* Patients can have unilateral, but not bilateral CNV. In the case of unilateral CNV, the eye without the CNV will be the study eye.
* Age greater than 50
* Willing and able to comply with clinic visit and study-related procedures
* Provide signed informed consent
* Able to understand and complete study-related questionnaire
* Be able to tolerate dilating drops

Exclusion Criteria:

* Bilateral CNV
* Other retinal degenerations and retinal vascular diseases such as diabetic retinopathy or macular edema, prior retinal surgery
* Pregnant, lactating, or currently expecting a child

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AMD with and without RMD
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-08-02 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
Proportion of CAD+ patients in RMD+ Patients | 6 months
  Rate of coronary artery disease in age-related macular disease patients with reticular macular disease
Proportion of CAD+ patients in RMD- Patients | 6 months
  Rate of coronary artery disease in age-related macular disease patients without reticular macular disease

SECONDARY OUTCOMES:
Evaluation of CAD risk factors as predictors of RMD status | 6 months
  Investigating the relationship between AMD/RMD to cardiac risk factors such as tobacco use, hyperlipidemia, elevated C-Reactive protein an inflammatory biomarker, and hypertension.
Correlation of lipid panels with RMD status | 6 months
  Measuring the total cholesterol in blood, the standard cholesterol test (called a "lipid panel") measures three specific kinds of fat: Low-density lipoproteins (LDL). High-density lipoproteins (HDL). Triglycerides.
Correlation of the C-Reactive Protein as an inflammatory biomarker with RMD status | 6 months
  High sensitivity CRP (hsCRP) blood tests able to measure down to 0.3 mg/L which is necessary in risk assessment for vascular disease.
Correlation of imaging features with RMD status | 6 months
  Correlation of presence of soft drusen, geographic atrophy or choroidal neovascularization status in fellow eye, if present, with RMD status
Correlation of genetic markers with CFHY402H and CFHrs1410996 genotypes, adjusting for AMD grade. These phenotypes may be a marker of genetic susceptibility for patients with RMD status. | 6 months
  High sensitivity RMD genetic blood test for markers with RMD status

CONTACTS AND LOCATIONS:
Overall Officials: R. Theodore Smith, MD PhD, Study Chair — New York Eye And Ear Infirmary of Mount Sinai
Locations (1):
- New York Eye and Ear Infirmary, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomson RJ, Chazaro J, Otero-Marquez O, Ledesma-Gil G, Tong Y, Coughlin AC, Teibel ZR, Alauddin S, Tai K, Lloyd H, Scolaro M, Govindaiah A, Bhuiyan A, Dhamoon MS, Deobhakta A, Narula J, Rosen RB, Yannuzzi LA, Freund KB, Smith RT. SUBRETINAL DRUSENOID DEPOSITS AND SOFT DRUSEN: Are They Markers for Distinct Retinal Diseases? Retina. 2022 Jul 1;42(7):1311-1318. doi: 10.1097/IAE.0000000000003460. PMID 35213528